CLINICAL TRIAL: NCT03945422
Title: The Use of Radio Frequency in Premature Jowl and Neck Laxity Following Facialplasty
Brief Title: The Use of RF in Premature Jowl and Neck Laxity Following Facialplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO608522A
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Premature Jowl and Neck Laxity Following Facialplasty

STUDY DESIGN:
Intervention Model Description: Subjects will receive the treatment and outcome will be followed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Subject will receive AccuTite/FaceTite and Morpheus8 treatment
  Interventions: Device: AccuTite/FaceTite

INTERVENTIONS:
Device: AccuTite/FaceTite — Radiofrequency-assisted lipolysis (RFAL) Morpheus8: Fractional RF
  Other Names: Morpheus8

SUMMARY:
Study is to evaluate the efficacy of treatment Radio Frequency in premature jowl and neck laxity following facialplasty

ELIGIBILITY:
Inclusion Criteria:

* Adult females and males between the ages of 40-80 inclusive, having premature jowl and/or neck laxity one to fifteen years following facialplasty, seeking skin tightening treatments.
* Lack lipodystrophy in the jowl or neck area or at least not amenable to liposuction improvement (not a candidate for liposuction).
* Lack of previous Face Lift complications (no nerve injury or hematoma history).
* The patients should understand the information provided about the investigative nature of the treatment, possible benefits and side effects, and sign the Informed Consent Form, (including thepermission to use photography).
* The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other aesthetic treatment methods for the last 6 months and during the entire study period.

Exclusion Criteria:

* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* The Handpiece should be used at least 1cm away from cochlear implants in the ear.
* Superficial permanent implant in the treated area such as metal plates and screws, metal piercing, silicone implants or an injected chemical substance.
* Current or history of skin cancer (remission of 5 years), or current condition of any other type of cancer, or pre-malignant moles.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy and nursing.
* History of bleeding coagulopathies or use of anticoagulants
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV or use of immunosuppressive medications.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction and hormonalvirilization.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* Any surgery or treatment such as laser or chemicals in treated area within 3-6 months prior to treatment or before complete healing.
* Allergies, in particular to anesthesia.
* Mental disorders such as Body Dysmorphic Disorder (BDD).
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Change in skin appearance | 3 months, 6 month, 9 months
  Photos from all time points (baseline and follow-up visits) will be evaluated by the treating physician and 2 independent evaluators.

SECONDARY OUTCOMES:
Investigator assessment of the skin appearance | 3 Month, 6 Months, 9 Months
  Investigator assessment of the skin appearance improvement comparing pre and post treatment using 0 - 4 -points Likert scale: 4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement ; 0 = No difference.
Optional: 3D Photographic analysis | 3 months, 6 month, 9 months
  3D Photographic analysis will be conducted using QuantifiCare System
Evaluate changes in skin appearance comparing photographs using Mechanical Turk (MTurk). The pictures will be sent through the system and evaluated by crowd workers. | 3 Months, 6 Months
  The pictures will be sent through the system and evaluated by crowd workers.

CONTACTS AND LOCATIONS:
Locations (1):
- Chicago Center for Facial Plastics, Chicago, Illinois, United States